CLINICAL TRIAL: NCT01582230
Title: A 24-week, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Vildagliptin 50mg Bid as an add-on Therapy to Insulin, With or Without Metformin, in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Vildagliptin 50mg Bid as an add-on Therapy to Insulin With or Without Metformin, in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A23155
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (Experimental): Eligible patients will receive vildagliptin 50 mg in addition to their stable dose of insulin with or without metformin. One tablet should be taken twice daily as one tablet before breakfast meal and one tablet before the evening meal for 24 weeks.
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator): Eligible patients will receive matching placebo in addition to their stable dose of insulin with or without metformin. One tablet should be taken twice daily as one tablet before breakfast meal and one tablet before the evening meal for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — Patient will receive vildagliptin 50mg twice daily (bid) in addition to their stable dose of insulin with or without metformin for 24 weeks
  Other Names: Galvus, LAF237
  Arms: Vildagliptin
Drug: Placebo — Patient will receive matching placebo to vildagliptin in addition to their stable dose of insulin with or without metformin for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of vildagliptin 50mg bid add-on therapy to improve overall glycemic control in patients with type 2 diabetes mellitus inadequately controlled on insulin with or without metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of Type2 diabetes mellitus (T2DM) by standard criteria
* C-peptide >0.6 ng/ml (>0.20 nmol/L).
* HbA1c ≥7.5 to ≤11% at Visit 1
* Treatment with stable, once or twice daily doses (maximum dose of < 1 unit/kg/day) of basal (long-acting, intermediate-acting) insulin alone or pre-mixed insulin for at least 12 weeks prior to Visit 1. Stable is defined as ±10% of the Visit 1 dose during the previous 12 weeks
* Patients receiving metformin must be on a stable dose of metformin (at least 1500 mg daily or a maximally tolerated dose) for at least 12 weeks prior to Visit 1
* Body Mass Index (BMI) ≥20 to ≤40 kg/m2 at Visit

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for participation in the study

* Fasting plasma glucose (FPG) ≥240 mg/dl (13.3 mmol/L) at Visit 1
* Pregnant or lactating women
* Acute metabolic diabetes complications such as ketoacidosis or hyperosmolar state (coma) within the past 6 months
* Current diagnosis of congestive heart failure (NYHA III or IV).
* Myocardial infarction (MI) within the past 6 months
* Liver disease such as cirrhosis or chronic active hepatitis

Other protocol defined inclusion/excusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin (HbA1c) at study endpoint, assessed in overall study population | Baseline and every study visit up to 24 weeks
  HbA1c analysis will be performed on a blood sample obtained by study personnel at every visit and measured by ion exchange HPLC. Study endpoint is defined as final available post- randomization assessment obtained at any visit prior to or at the start of major change in insulin use, up to final scheduled study visit (week 24 visit) inclusive.
Change from baseline in glycosylated hemoglobin (HbA1c) at study endpoint, assessed in Chinese study population | Baseline and every study visit up to 24 weeks
  HbA1c analysis will be performed on a blood sample obtained by study personnel at every visit and measured by ion exchange HPLC. Study endpoint is defined as final available post- randomization assessment obtained at any visit prior to or at the start of major change in insulin use, up to final scheduled study visit (week 24 visit) inclusive.

SECONDARY OUTCOMES:
Number of patients with adverse events, serious adverse events and death on over all population | 24 weeks
  Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Change from baseline after 24 weeks of treatment in fasting plasma glucose (FPG)on overall population | Baseline, week 24
  FPG will be performed on the blood samples collected at all every study visits from baseline to week 24.
Percentage of patients meeting responder criteria after 24 weeks treatment on overall population | After 24 weeks
  Responder rate will be analyzed in the following categories:
  * Endpoint HbA1c ≤ 6.5%
  * Endpoint HbA1c < 7%
  * Endpoint HbA1c <7% in patients with baseline HbA1c ≤ 8% The percentage of patients meeting each of the responder criteria as described, as well as the percentage of patients meeting any of these criteria in each treatment group will be computed
Number of patients with adverse events, serious adverse events and death on Chinese population | 24 weeks
  Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Change from baseline after 24 weeks of treatment in fasting plasma glucose (FPG) on Chinese population | Baseline, week 24
  FPG will be performed on the blood samples collected at all every study visits from baseline to week 24.
Percentage of patients meeting responder criteria after 24 weeks treatment on Chinese population | After 24 weeks
  Responder rate will be analyzed in the following categories: • Endpoint HbA1c ≤ 6.5% • Endpoint HbA1c < 7% • Endpoint HbA1c <7% in patients with baseline HbA1c ≤ 8% The percentage of patients meeting each of the responder criteria as described, as well as the percentage of patients meeting any of these criteria in each treatment group will be computed

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- China (12):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Philippines (3):
  - Novartis Investigative Site, Pasay, Philippines
  - Novartis Investigative Site, Metro Manila
  - Novartis Investigative Site, Quezon City
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- Thailand (3):
  - Novartis Investigative Site, Bangkok, Bangkok
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Khon Kaen

REFERENCES:
- [Derived] Ning G, Wang W, Li L, Ma J, Lv X, Yang M, Wang W, Woloschak M, Lukashevich V, Kothny W. Vildagliptin as add-on therapy to insulin improves glycemic control without increasing risk of hypoglycemia in Asian, predominantly Chinese, patients with type 2 diabetes mellitus. J Diabetes. 2016 May;8(3):345-53. doi: 10.1111/1753-0407.12303. PMID 25929739